CLINICAL TRIAL: NCT01433900
Title: The Advantage of Switching From Preserved to Preserved-free Treatments in Glaucoma. A Clinical and Confocal Study.
Brief Title: Switching From Preserved to Preserved-free Treatments for Glaucoma.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Paolo Fogagnolo (Other)
Responsible Party: Sponsor-Investigator, Paolo Fogagnolo, Prof. Luca Rossetti, University of Milan
Organization: University of Milan (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSD-007
Record Dates: First submitted 2011-07-25; First posted 2011-09-14 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2011-09

CONDITIONS: Glaucoma
Keywords: glaucoma; intraocular pressure; ocular surface; benzalkonium chloride
MeSH Terms: conditions — Glaucoma | interventions — tafluprost; Latanoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tafluprost (Active Comparator): 1 drop of tafluprost to eligible eye(s) once daily (at 9 pm)
  Interventions: Drug: Tafluprost
- Latanoprost (Active Comparator): 1 drop of latanoprost to eligible eye(s) once daily (at 9 pm)
  Interventions: Drug: Latanoprost

INTERVENTIONS:
Drug: Tafluprost — 1 drop of tafluprost to eligible eye(s) once daily (at 9 pm)
  Arms: Tafluprost
Drug: Latanoprost — 1 drop of tafluprost to eligible eye(s) once daily (at 9 pm)
  Arms: Latanoprost

SUMMARY:
A 1-year prospective, randomized, investigator-masked trial comparing the confocal and clinical effects of treatment with unpreserved prostaglandins (tafluprost) versus preserved prostaglandins (latanoprost) in newly-diagnosed glaucoma patients.

DETAILED DESCRIPTION:
The study protocol comprises 5 visits: baseline, month 3, month 6, month 9, month 12.

At baseline a clinical evaluator will perform a complete ophthalmologic evaluation to confirm diagnosis. The following examinations will be done in the following sequence: anterior segment examination, Shirmer test, Break-up time test. Thereafter, a confocal evaluator will perform confocal microscopy of the central and the peripheral cornea. Finally, contact measurements will be done in the following order: IOP (which will be measured at 3 pm), pachimetry (only at baseline visit) and gonioscony (only at baseline visit). A 15 minutes interval will elapse between two consecutive tests.

ELIGIBILITY:
Inclusion Criteria:

* The patient is suffering from ocular hypertension, POAG, PEX, NTG. Glaucoma definition is based on the European Glaucoma Society Guidelines.
* The patient is newly-diagnosed
* No fluorescein staining at baseline and no observable signs of ocular surface disease
* No treatment with topical BAK-containing products for at least 6 months
* Treatment of naïve patients

Exclusion Criteria:

* Unwilling to sign informed consent
* Not at least 18 years old
* Ocular condition that are of safety concern and that can interfere with the study results
* Closed/barely open anterior chamber angles or history of acute angle closure.
* Ocular surgery or argon laser trabeculoplasty within the last year. Ocular inflammation/infection occurring within three months prior to pre-trial visit.
* Presence of the following ocular conditions: KCS, moderate-severe blepharitis, Rosacea, Sjogren syndrome, pterygium, contact lens users.
* Use of concomitant topical ocular medication that can interfere with study medication
* Hypersensitivity to benzalkonium chloride or to any other component of the trial drug solutions.
* Any corneal pathology
* Diabetes at any stage
* Other abnormal condition or symptom preventing the patient from entering the trial, according to the Investigator's judgement.
* Refractive surgery patients
* Women who are pregnant, are of childbearing potential and are not using adequate contraception or are nursing.
* Inability to adhere to treatment/visit plan.
* Have participated in any other clinical trial (i.e., requiring informed consent) within one to three month prior to pre-trial visit (depending on ethics committee decisions).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Changes in the difference in the fiber density of the subbasal nerves in the central cornea and in each of 4 limbal quadrants | Month 3, 6, 9, 12

SECONDARY OUTCOMES:
Changes in sub-basal nerve characteristics (reflectivity, beading, tortuosity) | Months 3, 6, 9 ,12
Changes in density of epithelial cells, Langerhans cells, endothelial cells | Month 3, 6, 9 ,12
Changes in ocular surface (symptom and sign scales, break-up time, Schirmer test) | Month 3, 6, 9, 12

CONTACTS AND LOCATIONS:
Overall Officials: Luca Rossetti, MD, Principal Investigator — San Paolo Hospital, Milan, Italy
Locations (1):
- San Paolo Hospital, Milan, Italy

REFERENCES:
- [Derived] Fogagnolo P, Dipinto A, Vanzulli E, Maggiolo E, De Cilla' S, Autelitano A, Rossetti L. A 1-year randomized study of the clinical and confocal effects of tafluprost and latanoprost in newly diagnosed glaucoma patients. Adv Ther. 2015 Apr;32(4):356-69. doi: 10.1007/s12325-015-0205-5. Epub 2015 Apr 19. PMID 25893514